CLINICAL TRIAL: NCT06525103
Title: Pulsed Electromagnetic Therapy Versus Whole Body Vibration on Quadriceps Strength Post Burn
Brief Title: PEMT Versus WBV on Quadriceps Strength Post Burn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Talaat Moustafa Moustafa, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEMT VS WBV on Qadri
Record Dates: First submitted 2024-07-02; First posted 2024-07-29 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Burns of Thigh

STUDY DESIGN:
Intervention Model Description: Thirty patients (male and female) who suffering from second degree burn with burned body surface area 10% _25% BSA will participate in this study, they will be recruited from Al-Ahrar Teaching Hospital at Alsharqiya Governorate, Egypt. Their ages will be ranged from 25 to 40 years
Who Masked: Participant
Masking Description: Thirty patients (male and female) who suffering from second degree burn with burned body surface area 10% _25% BSA will participate in this study, they will be recruited from Al-Ahrar Teaching Hospital at Alsharqiya Governorate, Egypt. Their ages will be ranged from 25 to 40 years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A): Fifteen patients will receive whole body vibration (Experimental)
  Interventions: Device: whole body vibration
- Group (B): Fifteen patients will receive pulsed electromagnetic field (PEMF) (Experimental)
  Interventions: Device: electromagnitic field therapy

INTERVENTIONS:
Device: electromagnitic field therapy — EMSCULPT device (BTL Industries Inc., Boston, MA) based on HIFEM technology.
  * Frequency : 50 or 60 Hz.
  * Intenisty: 0-100 .Input voltage: 230 V
  Arms: Group (B): Fifteen patients will receive pulsed electromagnetic field (PEMF)
Device: whole body vibration — Crazy fit machine.
  * Input voltage:220 V.
  * Frequency : 30 Hz.
  * Maximum power: 1500W.
  * Intensity:1 to 50 levels.
  Arms: Group (A): Fifteen patients will receive whole body vibration

SUMMARY:
The purpose of the study is to evaluate which is more effective pulsed electromagnetic field therapy or whole-body vibration on quadriceps strength after chronic burn.

DETAILED DESCRIPTION:
A burn is an injury to the skin or other organic tissue primarily caused by heat, radiation or radioactivity, electricity, friction, or contact with chemicals. It is the fourth most common type of trauma worldwide and a major cause of mortality and disability in developing countries. Patients with ≥ 20% total burn surface area (TBSA) injury are potentially predisposed to significant morbidity and mortality. The immobilization period after burn is accompanied by numerous detrimental effect namely sever deconditioning such as sever weakness, impaired motor control decrease cognitive status, pain, risk of graft shearing and psychological factors. Severe burns are typically followed by a hypermetabolic response that lasts for at least 9-12 months post-injury. The endocrine status is also markedly altered with an initial and then sustained increase in proinflammatory 'stress' hormones such as cortisol and other glucocorticoids, and catecholamines including epinephrine and norepinephrine by the adrenal medulla and cortex. These hormones exert catabolic effects leading to muscle wasting . Pulsed electromagnetic fields (PEMFs) are known to be a noninvasive, safe and effective therapy agent without apparent side effects. Numerous studies have shown that PEMFs possess the potential to become a stand-alone or adjunctive treatment modality for treating musculoskeletal disorders. There are emerging evidences showing that pulsed electromagnetic field (PEMF) can modulate mitochondrial activities for muscle gain. PEMF exposure on top of regular exercise training may promote muscle regeneration and tissue healing. Whole Body Vibration Training (WBVT) can be described as exercising on a platform with an oscillating motion. Whole Body Vibration (WBV) is a newly developed neuromuscular training method, in which vibrations of various frequencies are provided to mechanically stimulate the receptors in the body such as muscle spindles. Whole Body Vibration Training (WBVT) elicits a biological adaptation that is connected to the neural potentiation effect. In this effect the proprioceptive pathways are strongly stimulated by the vibration which results in reflexive muscle contractions. Although WBVT combined with resistance training is becoming increasingly popular in various training recommendations, there is still an ongoing debate in literature, whether there are additional effects of WBV on muscle fitness and muscle performance in comparison to conventional exercise.

ELIGIBILITY:
Inclusion Criteria:

* • Both sexes.

  * Their ages were ranged from 25 to 40 years.
  * Had second degree burn of 10 % to 25 %.
  * Their body mass index (BMI) was not exceeded 34.9 Kg/m2.
  * All patients were clinically and medically stable when attending the study

Exclusion Criteria:

* • Unstable cardiovascular problems like arrhythmia and heart failure.

  * Diabetes mellitus.
  * Chronic chest disease.
  * Patients on medications affecting muscle power as steroids.
  * Auditory and visual problems.
  * Pregnancy & lactation.
  * Patients with history of epilepsy.
  * Clinically significant peripheral vascular disease.
  * Musculoskeletal or neurological limitation to physical exercise.
  * Any cognitive impairment that interferes with prescribed exercise procedures.
  * Amputation of lower limb.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-18 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
measure the strengh of quadriceps | basline
  evaluate which is more effective pulsed electromagnetic field therapy or whole-body vibration on quadriceps strength after chronic burn

REFERENCES:
- [Background] Cheing GL, Li X, Huang L, Kwan RL, Cheung KK. Pulsed electromagnetic fields (PEMF) promote early wound healing and myofibroblast proliferation in diabetic rats. Bioelectromagnetics. 2014 Apr;35(3):161-9. doi: 10.1002/bem.21832. Epub 2014 Jan 3. PMID 24395219